CLINICAL TRIAL: NCT01296035
Title: A Phase II Evaluation of Panitumumab and Gemcitabine as Treatment for Women With Recurrent Epithelial Ovarian Cancer.
Brief Title: Panitumumab and Gemcitabine in Relapsed Ovarian Cancer
Acronym: PanGem
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Newer technologies available; poor accrual to study.
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Carolyn McCourt, Dr. Carolyn McCourt, Women and Infants Hospital of Rhode Island
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WIH 20050782
Record Dates: First submitted 2011-02-09; First posted 2011-02-15 (Estimated); Results first posted 2015-08-25 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-07

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: recurrent ovarian cancer; platinum-refractory ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Panitumumab and Gemcitabine (Experimental): Panitumumab and Gemcitabine
  Interventions: Biological: Panitumumab

INTERVENTIONS:
Biological: Panitumumab — Panitumumab 2.5 mg/kg on D1, D8, D15, and D22 and Gemcitabine 800 mg/m2 on D1, D8, and D15 of each 28 day cycle.

SUMMARY:
This is a study to find out if the study drug, panitumumab, when given with gemcitabine works in treating ovarian cancer and to find out what side effects occur when they are given together.

DETAILED DESCRIPTION:
Epithelial ovarian cancer (EOC) remains a leading cause of gynecologic cancer mortality in women, with more than 22,000 deaths per year in the United States alone. Due to the lack of effective screening strategies and subtle early symptoms, eighty percent of newly diagnosed patients have disease that is advanced. Despite cytoreductive surgery and adjuvant paclitaxel-based and platinum-based chemotherapy, 5-year survival rates continue to be less than 40%. For patients who become resistant to the platinum compounds (defined as progressive disease while on a platinum-based chemotherapy regimen (refractory) or within 6 months of completing a platinum-based chemotherapy regimen (resistant)),the outlook is particularly poor, and often heralds multi-drug resistant disease.

At the present time, the management of ovarian cancer in the platinum refractory disease state is limited to palliative intent. Patients with advanced, bulky tumors, poor performance status and nutritional compromise are unlikely to respond to therapy and may be best served by supportive care. The clinical management of refractory disease requires both patience and persistence. A patient with platinum refractory disease is begun on one of the agents with activity and an evaluation of response is made every 6-8 weeks of therapy. As long as the patient shows no signs of disease progression, the therapy can be continued unless there is unacceptable toxicity. When progressive disease is observed, another of the list of available agents can be used. It is likely that patients will receive multiple single agents during the chronic phase of their illness. Every effort should be made to balance disease response with toxicity and quality of life.

Based on this rational, this trial will be conducted to evaluate the safety and efficacy of panitumumab, a human antibody targeted to the EGF-R, and Gemcitabine, in treating women with recurrent platinum-refractory/resistant EOC. Our aim is to determine the safety and feasibility of gemcitabine and panitumumab therapy in this population and once completed, to proceed with an efficacy study using an expanded cohort.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of metastatic, advanced, or recurrent platinum-resistant epithelial ovarian, primary peritoneal or fallopian tube cancer.
* Prior first line therapy with a platinum and taxane based combination as adjuvant therapy
* Measurable disease defined by RECIST criteria
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* age > 18
* Karnofsky performance status > 70
* Up to three prior lines of cytotoxic therapy in the setting of recurrent disease.
* Estimated life expectancy of at least 3 months
* Women of child-bearing potential must have a negative pregnancy test
* Adequate hematopoietic function defined as:

  * ANC ≥ 1500/mm3
  * Platelets ≥ 100,000/mm3
  * Hemoglobin ≥ 9 g/dL
  * Magnesium ≥ lower limit of normal
  * Calcium ≥ lower limit of normal
* Adequate renal and hepatic function defined as:

  * Bilirubin ≤ 1.5 times upper limit of normal (ULN)
  * SGOT ≤ 3 times ULN
  * Alanine aminotransferase (ALT) ≤3xULN (if liver metastases ≤5xULN)
  * Alkaline phosphatase ≤ 3 times ULN
  * Creatinine ≤ 1.5 mg/dL times ULN
  * Creatinine clearance ≤ 50 mL/min

Exclusion Criteria:

* Prior anti-EGFr antibody therapy (e.g., cetuximab) or treatment with small molecule EGFr inhibitors (e.g., gefitinib, erlotinib, lapatinib)
* Prior treatment with gemcitabine
* Radiotherapy ≤ 14 days prior to enrollment.
* More than three lines of systemic chemotherapy for recurrent or advanced disease. Prior hormonal therapy is allowed.
* Prior immunotherapy, or experimental or approved proteins/antibodies
* Female subject is pregnant or breast-feeding.
* Patient has received other investigational drugs within 28 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Prior treatment with panitumumab
* Concurrent uncontrolled illness
* Ongoing or active infection
* History or active secondary cancer within the last 5 years, except for superficial basal cell skin cancers, curatively resected non-melanoma skin cancer
* Psychiatric illness or social situation that would preclude study compliance.
* History or known presence of central nervous system (CNS) metastasis
* Subjects requiring chronic use of immunosuppressive agents (e.g., methotrexate, cyclosporine)
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) < 1 year before randomization
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or any evidence of interstitial lung disease on baseline chest CT scan
* Known positive test(s) for human immunodeficiency virus infection, hepatitis C virus, acute or chronic active hepatitis B infection
* Major surgery within 28 days or minor surgery within 14 days of study enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-02; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn McCourt, MD, Principal Investigator — Women & Infants' Hospital
Locations (1):
- Women & Infants' Hospital, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Panitumuab and Gemcitabine: Panitumumab: Panitumumab 2.5 mg/kg on D1, D8, D15, and D22 and Gemcitabine 800 mg/m2 on D1, D8, and D15 of each 28 day cycle.
Period: Overall Study
Arm/Group | Panitumuab and Gemcitabine
Started | 8
Completed | 7
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Panitumuab and Gemcitabine
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate, Measured by RECIST Criteria
Description: Documentation of known measurable or evaluable disease parameters after every 2 cycles of treatment. If any patient is withdrawn for the study prior to completion of therapy a repeat evaluation will be done at that time.
Time Frame: Every 8 weeks while on-study
Population: Due to the small number of participants, data were not collected as planned
Arm/Group | Panitumuab and Gemcitabine
Number analyzed (Participants) | 0

2. Secondary Outcome: Adverse Events, Measured by Active Version of the NCI Common Toxicity Criteria
Description: Adverse events (AEs) will be recorded during the duration of the trial, whether or not the events are considered related to medication. All AEs considered to be related to trial therapy will be followed for resolution, including into the post-treatment period.
Time Frame: Every 4 weeks while on-study, up to 24 weeks
Population: Please see results section. In short, there were 3 serious adverse events (1 thromboembolic, 1 hypomagnesemia, 1 bowel obstruction). Additional adverse events included (in decreasing order) rash, fatigue, anemia, edema, thrombocytopenia, abdominal pain, epistaxis, hypocalcemia, and calciphylaxis
Measure: Number; unit: participants
Units Other Than Participants: events
Arm/Group | Panitumuab and Gemcitabine
Number analyzed (Participants) | 8
Number analyzed (events) | 33
participants | 8

ADVERSE EVENTS:
Arm/Group | Panitumuab and Gemcitabine
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panitumuab and Gemcitabine (N=8)
Thromboembolic event (Vascular disorders) | 1 (1)
Hypomagnesemia (Investigations) | 1 (2)
Bowel obstruction (Gastrointestinal disorders) | 1 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panitumuab and Gemcitabine (N=8)
Rash (Skin and subcutaneous tissue disorders) | 6 (6)
Platelet count decreased (Investigations) | 3 (4)
Fatigue (General disorders) | 6 (6)
Anemia (Investigations) | 5 (5)
Hypocalcemia (Investigations) | 1 (1)
Abdominal pain (General disorders) | 2 (2)
Epistaxis (General disorders) | 2 (2)
Edema-limbs (Skin and subcutaneous tissue disorders) | 3 (3)
Calciphylaxis (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated prematurely due to poor accrual. The outcome measures could not be analyzed due to the small number or participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No